CLINICAL TRIAL: NCT02012426
Title: The Effect of a Multi-component Weight Management Program on Appetite, Food Preference and Body Weight
Acronym: SWSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Principal Investigator, University of Leeds
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LDS-2013-SLW; KRISTAL No. (Other: RG.PSYC.100944)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Overweight; Obesity; Sedentary Lifestlye
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Participants enrolled in commercial weight management program
  Interventions: Behavioral: Weight management program
- Control group (Active Comparator): Participants enrolled in standard care weight management provision
  Interventions: Behavioral: Weight management program

INTERVENTIONS:
Behavioral: Weight management program

SUMMARY:
The aim of the current study is to demonstrate that a commercial weight management diet (i.e. low energy density) influences satiation, hunger and satiety and leads to lower energy intake during ad-libitum meals and over a full day. We further seek to demonstrate the sustainability of this effect following 12- week weight loss on the weight management program.

* We hypothesise that formulated (low energy) meals will lead to decreased hunger, greater fullness and reduced desire to eat compared to standard meals.
* We hypothesise that the commercial weight management program will lead to greater weight loss compared to control program.
* We hypothesise that formulated meals (high consumer acceptance) will improve hedonic control over eating (lower wanting for high fat food)
* We hypothesise that the commercial weight management program will improve hedonic control over eating (reduced experience food cravings)

ELIGIBILITY:
Inclusion Criteria:

* BMI of 28 - 45 kg/m2
* Reporting an interest in weight loss, not actively participating in a commercial weight loss program,
* Not increased physical activity levels in the past 2-4 weeks
* Able to eat most everyday foods and fruits and vegetables
* Written informed consent to be given

Exclusion Criteria:

* Significant health problems that could cause confounding effects between intervention and control.
* Taking any medication or supplements known to affect appetite or weight within the past month and/or during the study
* Pregnant, planning to become pregnant or breastfeeding
* History of anaphylaxis to food
* Known food allergies or food intolerance
* Smokers and those who have recently ceased smoking
* Participants receiving systemic or local treatment likely to interfere with evaluation of the study parameters
* Those who have previously taken part in a commercial weight loss program in the last 6 months? .
* Participants who work in appetite or feeding related areas
* Participants unable to consume foods used in the study
* Participants who have had bariatric surgery
* Participants with a history of eating disorder
* Presence of untreated hypothyroidism
* Inability to fully comply with intervention or study procedures
* Insufficient English language skills to complete study questionnaires

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Test Meal Energy Intake | Week 0 and week 12
  Measured reductions in ad-libitum energy intake following consumption of formulated test meal in comparison to control.
24h Energy Intake | Week 0 and week 12
  Measured reduction in total within-day energy intake following consumption of formulated meals in comparison to control
Appetite sensations | Week 0 and week 14
  Measured reduction in hunger and increase in satiety quotient following consumption of formulated test meal in comparison to equi-energetic control
Food preference | Week 0 and week 14
  Measured changes in food preference and liking and wanting profiles for food (HF<LF) following consumption of formulated test meal in comparison to equi-energetic control

SECONDARY OUTCOMES:
Body Weight | Weekly from week 0 to week 12
  Measured change in weight and energy balance parameters over a 12 week period following participation in commercial weight management program compared to control group.

OTHER OUTCOMES:
Food diary | Week 0 and week 12
  Intervention adherence and compensation through 1) food diary analysis.
Accelerometer | Week 0 and week 12
  Intervention adherence and compensation through accelerometer analysis.
Interview | Week 12
  Detailed feedback on participant experience of commercial weight management program through qualitative interview and marketing survey.

CONTACTS AND LOCATIONS:
Overall Officials: Graham S Finlayson, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Buckland NJ, Camidge D, Croden F, Myers A, Lavin JH, Stubbs RJ, Blundell JE, Finlayson G. Women with a low-satiety phenotype show impaired appetite control and greater resistance to weight loss. Br J Nutr. 2019 Oct 28;122(8):951-959. doi: 10.1017/S000711451900179X. PMID 31340872
- [Derived] Buckland NJ, Camidge D, Croden F, Lavin JH, Stubbs RJ, Hetherington MM, Blundell JE, Finlayson G. A Low Energy-Dense Diet in the Context of a Weight-Management Program Affects Appetite Control in Overweight and Obese Women. J Nutr. 2018 May 1;148(5):798-806. doi: 10.1093/jn/nxy041. PMID 30053284